CLINICAL TRIAL: NCT03197987
Title: Endocuff vs Transparent Cap To Increase Adenoma Detection Rate During Colonoscopy
Brief Title: Comparison of Two Devices During Colonoscopy
Acronym: COLONAUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, JAVIER SOLA VERA SANCHEZ, M.D, Ph D, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ADR-1
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Adenomatous Polyps
Keywords: adenoma detection rate; cap-assisted colonoscopy; endocuff
MeSH Terms: conditions — Adenomatous Polyps | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocuff colonoscopy (Experimental): Endocuff-assisted colonoscopy
  Interventions: Device: Endocuff
- Cap colonoscopy (Active Comparator): Cap-assisted colonoscopy
  Interventions: Device: cap

INTERVENTIONS:
Device: Endocuff — Endocuff-assisted colonoscopy
  Other Names: non
  Arms: Endocuff colonoscopy
Device: cap — Cap-assisted colonoscopy
  Other Names: non
  Arms: Cap colonoscopy

SUMMARY:
Colonoscopy is the gold standard investigation for the diagnosis of bowel pathology and colorectal cancer screening. Adenoma detection rate is a marker of high quality colonoscopy. In this study we compare two devices: Endocuff (TM) and cap that can increase the adenoma detection rate during colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard investigation for the diagnosis of bowel pathology and colorectal cancer screening. Adenoma detection rate is a marker of high quality colonoscopy and a high adenoma detection rate is associated with a lower incidence of interval cancers. Several technological advancements have been explored to improve adenoma detection rate. Endocuff Vision™ has been shown to improve adenoma detection rate in several studies. Cap-assisted colonoscopy is a technique that allow improved visualization of the colonic folds by flattening the fold within the viewing field. However, studies have reported mixed results on adenoma detection in cap-assisted colonoscopy.

This is a prospective, single-centre, randomized controlled trial comparing the adenoma detection rate in patients undergoing Endocuff Vision™-assisted colonoscopy versus cap-assisted colonoscopy. Patients are randomized according to bowel cancer screening status to receive Endocuff Vision™-assisted colonoscopy or cap colonoscopy on the day of procedure. Baseline data, colonoscopy, and polyp data including histology are collected. Patients are followed up at 30 days for complications. This study will take place in an University Hospital in Spain. A maximum of 9 expert colonoscopists will recruit a total of 712 patients.

This is the first trial to evaluate the adenoma detection rate of Endocuff Vision™ vs cap colonoscopy in all screening, surveillance, and diagnostic patient groups. This study will guide clinicians to decide what device to use to increase adenoma detection rate in routine colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* All patients who are attending for screening, surveillance or diagnostic colonoscopy.

Exclusion Criteria:

* patients with absolute contraindications to colonoscopy;
* patients with established or suspicion of large bowel obstruction or pseudo-obstruction;
* patients with known colonic strictures;
* patients with a known severe diverticular segment (that is likely to impede colonoscope passage);
* patients with active or known colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis);
* patients lacking capacity to give informed consent;
* patients on clopidogrel, warfarin, or other new generation anticoagulants who have not stopped this for the procedure;
* patients who are attending for a therapeutic procedure or assessment of a known lesion, or submitted for rectoscopy or rectosigmoidoscopy;
* examination performed by a non-expert colonoscopist;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 7 days
  number of patients with at least one adenoma/total number of patients

SECONDARY OUTCOMES:
mean adenoma per patient | 7 days
  total number of adenoma/total number of patient

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sola Vera, Ph.D., Principal Investigator — Hospital General Universitario de Elche
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] van Doorn SC, van der Vlugt M, Depla A, Wientjes CA, Mallant-Hent RC, Siersema PD, Tytgat K, Tuynman H, Kuiken SD, Houben G, Stokkers P, Moons L, Bossuyt P, Fockens P, Mundt MW, Dekker E. Adenoma detection with Endocuff colonoscopy versus conventional colonoscopy: a multicentre randomised controlled trial. Gut. 2017 Mar;66(3):438-445. doi: 10.1136/gutjnl-2015-310097. Epub 2015 Dec 16. PMID 26674360
- [Background] Marsano J, Tzimas D, Mckinley M, et al. Endocuff assisted colonoscopy increases adenoma detection rates: a multi-center study. Gastrointest Endosc 2014;79(5 Suppl):AB550
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Background] Horiuchi A, Nakayama Y, Kato N, Ichise Y, Kajiyama M, Tanaka N. Hood-assisted colonoscopy is more effective in detection of colorectal adenomas than narrow-band imaging. Clin Gastroenterol Hepatol. 2010 Apr;8(4):379-83. doi: 10.1016/j.cgh.2009.08.018. Epub 2009 Aug 26. PMID 19716434
- [Background] Rastogi A, Bansal A, Rao DS, Gupta N, Wani SB, Shipe T, Gaddam S, Singh V, Sharma P. Higher adenoma detection rates with cap-assisted colonoscopy: a randomised controlled trial. Gut. 2012 Mar;61(3):402-8. doi: 10.1136/gutjnl-2011-300187. Epub 2011 Oct 13. PMID 21997547
- [Background] Hewett DG, Rex DK. Cap-fitted colonoscopy: a randomized, tandem colonoscopy study of adenoma miss rates. Gastrointest Endosc. 2010 Oct;72(4):775-81. doi: 10.1016/j.gie.2010.04.030. Epub 2010 Jun 25. PMID 20579648
- [Background] Frieling T, Neuhaus F, Kuhlbusch-Zicklam R, Heise J, Kreysel C, Hulsdonk A, Blank M, Czypull M. Prospective and randomized study to evaluate the clinical impact of cap assisted colonoscopy (CAC). Z Gastroenterol. 2013 Dec;51(12):1383-8. doi: 10.1055/s-0033-1335637. Epub 2013 Dec 11. PMID 24338756
- [Background] de Wijkerslooth TR, Stoop EM, Bossuyt PM, Mathus-Vliegen EM, Dees J, Tytgat KM, van Leerdam ME, Fockens P, Kuipers EJ, Dekker E. Adenoma detection with cap-assisted colonoscopy versus regular colonoscopy: a randomised controlled trial. Gut. 2012 Oct;61(10):1426-34. doi: 10.1136/gutjnl-2011-301327. Epub 2011 Dec 20. PMID 22187070
- [Background] Morgan J, Thomas K, Lee-Robichaud H, Nelson RL. Transparent Cap Colonoscopy versus Standard Colonoscopy for Investigation of Gastrointestinal Tract Conditions. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD008211. doi: 10.1002/14651858.CD008211.pub2. PMID 21328306
- [Background] Pohl H, Bensen SP, Toor A, Gordon SR, Levy LC, Berk B, Anderson PB, Anderson JC, Rothstein RI, MacKenzie TA, Robertson DJ. Cap-assisted colonoscopy and detection of Adenomatous Polyps (CAP) study: a randomized trial. Endoscopy. 2015 Oct;47(10):891-7. doi: 10.1055/s-0034-1392261. Epub 2015 Jun 30. PMID 26126162
- [Derived] Sola-Vera J, Catala L, Uceda F, Pico MD, Perez Rabasco E, Saez J, Jimenez N, Arjona MD, Fernandez M, Girona E, Garcia-Sepulcre MF. Cuff-assisted versus cap-assisted colonoscopy for adenoma detection: results of a randomized study. Endoscopy. 2019 Aug;51(8):742-749. doi: 10.1055/a-0901-7306. Epub 2019 May 16. PMID 31096275